CLINICAL TRIAL: NCT03760614
Title: A Phase Ib Study of Entinostat and FOLFOX in Subjects With Pancreatic Adenocarcinoma
Brief Title: A Study of Entinostat and FOLFOX in Subjects With Pancreatic Adenocarcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19218
Record Dates: First submitted 2018-11-26; First posted 2018-11-30 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — entinostat; Folfox protocol

STUDY DESIGN:
Intervention Model Description: This will be a modified 3+3 dose-escalation design with a primary endpoint of dose-limiting toxicity. All cohorts will receive the same dose of FOLFOX, once every 2 weeks. All cohorts will receive entinostat on days 1,8, 15, and 22 of 28 day cycles. Cohorts will vary in their dose of entinostat as follows:
  * Cohort 0: 2mg
  * Cohort 1: 3mg
  * Cohort 2: 4mg
  * Cohort 3: 5mg
  Dosing will start with cohort 1. If no dose limiting toxicities (DLTs) are observed, the dose will be escalated directly to cohort 3. If any DLTs are experienced in cohort 1, three additional subjects will be enrolled in cohort 1. If no DLTs are experience by the additional subjects, the dose will be escalated to cohort 2. If a DLT occurs in two subjects in any dose cohort, dose escalation will be halted, and the next three subjects will be enrolled at the next lower dose cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entinostat + FOLFOX (Experimental): FOLFOX will be administered intravenously (IV), into a vein, using a port-a-cath every 2 weeks. Entinostat will be administered orally on days 1, 8, 15 and 22 of each 28-day cycle. Entinostat dose will vary between 2mg and 5mg depending on time of enrollment and observed toxicities. Dosing will begin at 3mg.
  Interventions: Drug: Entinostat; Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Entinostat — Entinostat will be administered orally on days 1, 8, 15 and 22 of each 28-day cycle.
Drug: FOLFOX regimen — FOLFOX will be administered intravenously (IV), into a vein, using a port-a-cath every 2 weeks.

SUMMARY:
The main purpose of this study is to find the best dose of entinostat when given in combination with FOLFOX for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Ability to comply with the protocol.
* Aged ≥ 18 years.
* Histologically or cytologically confirmed metastatic pancreatic adenocarcinoma that has progressed after first-line gemcitabine+nab-paclitaxel-based chemotherapy.
* ECOG PS of 0 or 1
* At least one lesion that can be measured accurately at baseline as ≥10mm in the longest diameter (except lymph nodes which must have a short axis ≥15mm) with CT/MRI and which is suitable for repeated measurements per RECIST v1.1
* Adequate hematological and end-organ function, as per the local institutions reference ranges, within 72 hrs prior to day 1 of cycle 1 of treatment defined by the following:

  1. Hematology: ANC ≥1.5 x 109/L (≥1500 cells / mm3); Platelet count ≥ 150 x 109/L (≥150,000 cells/mm3); Hb ≥ 9g/dl (≥9 mg/L)
  2. Coagulation: INR and aPTT ≤1.5 x ULN.
  3. Hepatic function: bilirubin ≤1.5 x ULN; AST / ALT ≤ 2.5 x ULN (or ≤ 5 x ULN in the presence of liver metastasis)
  4. Renal: Creatinine < 1.5x ULN or calculated creatinine clearance ≥ 50ml/min calculated as per local institution standards.
* Negative serum or urine pregnancy test within 14 days of day 1 cycle 1 for female subjects of childbearing potential. Female subjects of childbearing potential as well as male subjects must agree to use effective contraception during the study and for 120 days after the last of entinostat. Non-childbearing potential is defined as:

  1. ≥45 years of age and has not had menses for >2 years
  2. Amenorrhoeic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation
  3. Post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure otherwise the subject must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of study drug
* Tumor sites amenable to repeated biopsies.
* Willingness to undergo paired tumor biopsies during the trial.

Exclusion Criteria:

* Subjects with known or suspected brain metastasis
* Significant cardiovascular disease such as New York Heart Associate Class III/IV, cardiac failure, myocardial infarction within 6 months prior to enrolment, unstable arrhythmia, or evidence of ischemia on ECG.
* Baseline QTc exceeding 450msec (470msec for females) and / or subjects receiving class 1A or class III anti-arrhythmic agents.
* Known HIV or active hepatitis A, B or C infection (with positive viral PCR).
* Malignancies other than pancreatic cancer ≤5 years prior to Entinostat and FOLFOX cycle 1 day 1, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcomes (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of PSA relapse or incidental prostate cancer (Gleason score ≤3 +4 and PSA <10ng/L undergoing active surveillance and treatment naïve).
* Severe infections ≤ 4 weeks prior to enrolment in the study as well as active, uncontrolled bacterial, viral or fungal infections requiring systemic treatment.
* Major surgical procedure ≤ 2 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
* Treatment with chemotherapy or other investigational agents within 28 days (or at least 5 x the half-life of the drug) prior to day 1 cycle 1 of Entinostat and FOLFOX (6 weeks for nitrosoureas or Mitomycin C).
* Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational medicinal product (IMP) within ≤ 5 x the half-life of the IMP prior to day 1 cycle 1 of Entinostat and FOLFOX.
* Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of Entinostat or FOLFOX, may affect the interpretation of the results, render the subject at high risk from treatment complications or interferes with obtaining informed consent.
* Female subjects who are pregnant or nursing.
* Pre-existing neuropathy > CTCAE Grade 2
* Previous treatment with platinum agents
* Allergy to benzamide or inactive components of entinostat
* Any contraindication to oral agents or significant nausea and vomiting, malabsorption or significant small bowel resection that, in the opinion of the investigator, would preclude adequate absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | During the first 28 days of treatment
  Dose limiting toxicity (DLT)

SECONDARY OUTCOMES:
Incidence, nature and severity of adverse events (AE) | From time of enrollment until completion of the Safety Visit 30 days (+/- 7) days after last dose of entinostat (treatment with entinostat may continue until disease progression, death, unacceptable toxicites or withdrawal, estimated time 6 months)
  Incidence, nature and severity of adverse events (AE)
Progress free survival (PFS) | From study entry until disease progress or death from any cause, whichever occurs first (assessed at 6 months)
  Progress free survival (PFS)
Overall response rate (ORR) | Through study completion, estimated 1 year
  Overall response rate (ORR) as defined as proportion of patients with complete response (CR) or partial response (PR)

IPD SHARING:
Plan to Share IPD: Undecided